CLINICAL TRIAL: NCT02257710
Title: BIOTRONIK - SaFety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III United Kingdom Satellite
Brief Title: BIOFLOW-III UK Satellite Registry Orsiro Stent System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biotronik UK Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: G1402
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Diseases
Keywords: national; Multicenter; Observational registry; Orsiro Drug Eluting Stent (DES); Stenting; Treatment of coronary artery disease; Coronary revascularization; Coronary Intervention; STEMI; NSTEMI; Ischemia; Angina; Acute Myocardial Infarction (AMI); Small Vessels; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro: All subjects requiring coronary revascularization with Drug Eluting Stents (DES)
  Interventions: Device: Orsiro

INTERVENTIONS:
Device: Orsiro

SUMMARY:
Clinical evaluation of the Orsiro LESS in subjects requiring coronary revascularization with Drug Eluting Stents (DES). 500 subjects will be enrolled in this registry.

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD) treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedure success. However, the medium to long-term complications range from rather immediate elastic coil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30 to 50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in De Novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20 to 40% of cases, necessitating repeat procedures.

The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

Therefore this observational registry has been designed for the clinical evaluation of the ORSIRO LESS requiring coronary revascularization with DES. It is designed to investigate and collect clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in an all-comers patient population in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease
* Subject signed informed consent for data release
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject did not sign informed consent for data release
* Pregnancy
* Known intolerance to aspirin, clopidogrel, Ticlopidine, heparin or any other anticoagulant/antiplatelet therapy required for PCI, stainless steel, Sirolimus or contrast media
* Planned surgery within 6 months after PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint not reached yet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects from an all-comers patient population with all subjects requiring coronary revascularization with a Drug Eluting Stent (DES).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
TLF | 6 months
  Composite of cardiac death, target vessel Q-wave or non Q-wave Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG) and clinically driven Target Lesion Revascularization (TLR)
Target Vessel Revascularization (TVR) | 6 and 12 months
  Any repeat revascularization of the target vessel.
Target Lesion Revascularization (TLR) | 6 and 12 months
  Defined as any repeat revascularization of the target lesion.
Stent Thrombosis | 6 and 12 months
  Definite, Probable and Possible Stent Thrombosis
Clinical Device Success | up to seven days
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without use of a device outside the assigned treatment strategy.
Clinical Procedural success | up to seven days
  Successful delivery and deployment of the investigational stent (s) at the intended target lesion and successful withdrawal of the stent delivery system with attainment of a final residual stenosis of less than 50% by visual estimation and without using any adjunctive device without the occurrence of ischemia-driven major adverse cardiac event during the hospital stay to a maximum of the first seven days post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mahmoudi, MD, Principal Investigator — St. Peter's Hospital
Locations (4):
- United Kingdom (4):
  - Royal Sussex County Hospital, Brighton, East-Sussex
  - St Peter's Hospital, Chertsey, Surrey
  - University Hospital Southampton, Southampton
  - Royal Cornwall Hospital, Truro